CLINICAL TRIAL: NCT00777764
Title: The Safety and Utility of Skin Testing With XOLAIR® (Omalizumab) and Placebo Omalizumab (Formulation Excipients)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Q4465g
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Asthma
Keywords: Xolair; Asthma; Skin Tests
MeSH Terms: conditions — Asthma | interventions — KPNA1 protein, human

ARMS (2):
- Healthy Volunteers (Experimental): Healthy participants were tested sequentially in a skin prick test procedure with positive control (histamine 6 mg/mL), negative control (saline), and 1:1000, 1:100, 1:10 dilution and full concentrations of both omalizumab and omalizumab excipients.
  Interventions: Drug: Cohort I
- Allergic Asthma Participants (Experimental): Allergic asthma participants were tested sequentially in a skin prick test procedure with positive control (histamine 6 mg/mL), negative control (saline), and a succession of 1:1000, 1:100, 1:10 dilutions and full concentration of both omalizumab and omalizumab excipients.
  Interventions: Drug: Cohort 2

INTERVENTIONS:
Drug: Cohort I — In sterile water for injection (SWFI), full concentration and 1:1000, 1:100, 1:10 dilutions of 125 mg/mL of standard solution of omalizumab and its excipients. Skin prick test of each dilution concentration of 1:1000, 1:100, 1:10 and full concentration and Intradermal tests of each dilution concentration of 1:1000, 1:100 and 1:10 were followed by 20 minutes of observation. For the skin prick test, participants were tested initially with positive control (histamine 6 mg/mL) and negative control (saline), and with omalizumab and its excipients simultaneously from the lowest concentration.
  For the intradermal test, participants were tested initially with positive control (histamine 0.1 mg/mL) and negative control (saline), and with omalizumab and its excipients simultaneously from the lowest concentration.
  Dilutions of omalizumab and its excipients were in SWFI.
  Arms: Healthy Volunteers
Drug: Cohort 2 — In a saline solution, full concentration and 1:1000, 1:100, 1:10 dilutions of 125 mg/mL of standard solution of omalizumab and its excipients. Skin prick test of each dilution concentration of 1:1000, 1:100, 1:10 and full concentration and Intradermal tests of each dilution concentration of 1:100,000 and 1:10,000 were followed by 20 minutes of observation.
  For the skin prick test, participants were tested initially by positive control (histamine 6 mg/mL) and negative control (saline), and with omalizumab and its excipients simultaneously from the lowest concentration. For the intradermal test, participants were tested initially with positive control (histamine 0.1 mg/mL) and negative control (saline), and with omalizumab and its excipients simultaneously from the lowest concentration.
  Dilutions of omalizumab and its excipients were made in saline.
  Arms: Allergic Asthma Participants

SUMMARY:
This study enrolled 30 healthy volunteers and 30 patients with atopic asthma, for a total of 60 subjects. The study examined the tolerability of omalizumab and omalizumab excipients in two successive cohorts of subjects, healthy volunteers and patients with allergic asthma without prior exposure to omalizumab, according to a skin test protocol, consisting of a prick skin test and/or intradermal test.

ELIGIBILITY:
Inclusion Criteria:

* (Applicable to healthy subjects only) Healthy subjects not taking any regular prescription medication, without history of allergy, and considered healthy by the physician
* (Applicable to asthma patients only) Patients with atopic asthma diagnosed by a physician with asthma and history of positive skin test(s)
* Physical examination findings within normal limits
* Body mass index (BMI) between 18 and 30, inclusive

Exclusion Criteria:

* Pregnancy and lactation
* Current or previous treatment with a biologic agent (e.g., monoclonal antibody)
* Concurrent disease or condition that would interfere, or for which the treatment might interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to individuals in this study
* History or symptoms of significant psychiatric disease, including but not limited to, depression, schizophrenia, etc.
* History of drug abuse
* Participation in an investigational drug or device trial within the last 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wong, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects: Healthy participants were tested sequentially in a skin prick test procedure with positive control (histamine 6 mg/mL), negative control (saline), and 1:1000, 1:100, 1:10 dilution and full concentrations of both omalizumab and omalizumab excipients. Without reaction, this then followed a sequential intradermal test procedure with positive control (histamine 0.1 mg/mL), negative control (saline), and 1:1000, 1:100 and 1:10 dilution concentrations of omalizumab and its excipients. There was a 20 minute observation period following all dosings.
  Excipients include sucrose, histidine, histidine hydrochloride monohydrate and polysorbate 20.
  Dilutions of omalizumab and its excipients were made in sterile water for injection (SWFI).
- Allergic Asthma Participants: Allergic asthma participants were tested sequentially in a skin prick test procedure with positive control (histamine 6 mg/mL), negative control (saline), and a succession of 1:1000, 1:100, 1:10 dilutions and full concentration of both omalizumab and omalizumab excipients. Without reaction, this then followed a sequential intradermal test procedure with positive control (histamine 0.1 mg/mL), negative control (saline), and 1:100,000 and 1:10,000 dilution concentrations of omalizumab and its excipients. There was a 20 minute observation period following all dosings.
  Excipients include sucrose, histidine, histidine hydrochloride monohydrate and polysorbate 20.
  Dilutions of omalizumab and its excipients were made in saline solution.
Period: Overall Study
Arm/Group | Healthy Subjects | Allergic Asthma Participants
Started | 30 | 30
Completed | 30 | 29
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | Allergic Asthma Participants | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (13.10) | 32.0 (10.88) | 32.9 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 17 | 24
  Male | 23 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by of Adverse Events Following a Skin Test Procedure
Description: Skin test procedures were skin prick test or intradermal test. The test started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped. Subjects were observed for 20 minutes following each test; subjects were observed for 1 hour after the last intradermal test. Those with a positive response were observed for an additional 6 hours.
  Severity refers to the intensity of an AE (mild, moderate or severe). Mild is itching or hives, for example. A severe event requires emergency medical treatment and can result in death.
Time Frame: Up to 7 days following skin testing
Population: Safety population, defined as subjects who received at least one concentration of omalizumab or omalizumab excipient.
Measure: Number; unit: participants
Arm/Group | Healthy Subjects | Allergic Asthma Participants
Number analyzed (Participants) | 30 | 30
participants
  Any adverse event | 1 | 3
  Severity: Mild | 0 | 0
  Severity: Moderate | 1 | 3
  Severity: Severe | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced a Positive Skin Reaction (Skin Prick Test)
Description: For skin prick, positive control (histamine 6 mg/mL) and negative control (saline) were used. Positive skin reaction was defined as a ≥ 3-mm wheal and/or > 10-mm erythema from negative control. The skin prick test started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped.
Time Frame: on the day of skin test
Population: Safety population, defined as subjects who received at least one concentration of omalizumab or omalizumab excipient. For healthy volunteer cohort, undiluted: n=29. The skin tests started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped (i.e., reason for different Ns per dilution.)
Measure: Number; unit: participants
Arm/Group | Healthy Subjects | Allergic Asthma Participants
Number analyzed (Participants) | 30 | 30
participants
  1:1000 Dilution; Excipient | 0 | 0
  1:1000 Dilution; Omalizumab | 0 | 0
  1:100 Dilution; Excipient | 0 | 0
  1:100 Dilution; Omalizumab | 0 | 0
  1:10 Dilution; Excipient | 1 | 0
  1:10 Dilution; Omalizumab | 0 | 0
  Undiluted; Excipient | 2 | 0
  Undiluted; Omalizumab | 0 | 0

3. Primary Outcome: Number of Participants Who Experienced a Positive Skin Reaction (Intradermal Test in Healthy Volunteers)
Description: For intradermal testing, positive control (histamine 0.1 mg/mL) and negative control (saline) were used. Positive skin reaction was defined as a ≥ 3-mm wheal and/or > 10-mm erythema from negative control. The intradermal test started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped.
Time Frame: on the day of skin test
Population: Safety population. For 1:1000 dilutions: n=27; for 1:100 dilutions: n=21; for 1:10 dilutions: n=13. The skin tests started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped (i.e., reason for different Ns per dilution.)
Measure: Number; unit: participants
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 27
participants
  1:1000 Dilution; Excipient | 6
  1:1000 Dilution; Omalizumab | 2
  1:100 Dilution; Excipient | 7
  1:100 Dilution; Omalizumab | 6
  1:10 Dilution; Excipient | 0
  1:10 Dilution; Omalizumab | 0

4. Primary Outcome: Number of Participants Who Experienced a Positive Skin Reaction (Intradermal Test in Patients With Allergic Asthma)
Description: as for outcome 3
Time Frame: on the day of skin test
Population: Safety population. For 1:100,000 dilutions: n=30; for 1:10,000 dilutions: n=29. The skin tests started with the lowest concentration. If a positive skin reaction was observed, escalation to the next dilution was stopped (i.e., reason for different Ns per dilution.)
Measure: Number; unit: participants
Arm/Group | Patients With Allergic Asthma
Number analyzed (Participants) | 30
participants
  1:100,000 Dilution; Excipient | 1
  1:100,000 Dilution; Omalizumab | 0
  1:10,000 Dilution; Excipient | 4
  1:10,000 Dilution; Omalizumab | 7

ADVERSE EVENTS:
Description: Safety-evaluable population.
  Note: The incidence of each AE is reported as the number of participants experiencing the event, not the number of occurrences for each AE. AEs are reported regardless of the investigator's assessment of relation to study drug.
Arm/Group | Healthy Subjects | Allergic Asthma Participants
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Subjects (N=30) | Allergic Asthma Participants (N=30)
Gastroenteritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.